CLINICAL TRIAL: NCT05520554
Title: Development, Reliability and Validity of the Telerehabilitation Satisfaction Questionnaire- TrSQ in Neurological Diseases
Brief Title: Development, Reliability and Validity of the Telerehabilitation Satisfaction Questionnaire- TrSQ
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sefa Eldemir, Principal Investigator, Gazi University
Other Study IDs: 4- ND-Development-TSQ
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Neurological Disease
Keywords: Multiple Sclerosis; Parkinson Disease; Stroke; Telerehabilitation; Satisfaction
MeSH Terms: conditions — Nervous System Diseases; Multiple Sclerosis; Parkinson Disease; Stroke; Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telerehabilitation Satisfaction: Telerehabilitation Satisfaction Group
  Interventions: Other: Development of the Telerehabilitation Satisfaction Questionnaire

INTERVENTIONS:
Other: Development of the Telerehabilitation Satisfaction Questionnaire — This study will be examined the development, validity, and reliability of the Telerehabilitation Satisfaction Questionnaire in patients with MS.

SUMMARY:
Parkinson's disease (PD), stroke, and Multiple Sclerosis (MS) are the most common neurological diseases. Today, physiotherapy and rehabilitation approaches together with optimal medical and surgical treatment form the basis of treatment for these diseases. Recently, it has been stated that various telerehabilitation interventions in the field of physiotherapy and rehabilitation may be an additional option to the rehabilitation approaches applied in the clinic. In addition, there are benefits such as continuity in patient education and rehabilitation, saving time and expenditure of individuals on the road. However, some problems arise in this form of treatment. Especially weak internet connection, sometimes requiring technical knowledge and expensive equipment can reduce the participation and satisfaction level of individuals. It is also important to evaluate the level of satisfaction in expanding the usability of telerehabilitation services and determining the best telerehabilitation service. For this reason, there is a need for questionnaires investigating the satisfaction level of physiotherapy and rehabilitation applied through telerehabilitation.

DETAILED DESCRIPTION:
Questionnaire items were created in two stages. First, 5 experts will independently review the literature on "telerehabilitation" and "satisfaction". In addition, these experts will be asked to create a pool of questions based on their experiences in telerehabilitation and by taking the opinions of patients receiving telerehabilitation about satisfaction. Then, 5 experts will come together and obtain a single question pool containing the questions they deem important in their question pool. The second step will involve scaling the elements. In this study, scale items will be scored on a five-point Likert scale, ranging from 1, strongly disagree to 5, strongly agree.

Then, it will be applied to a pilot group of 10 people and it will be evaluated whether the items prepared by the experts are understood by the patients. In line with the expert opinion and the result of the pilot study, the final version of the scale will be decided and applied to MS, PD, and stroke patients who make up the study group. Finally, the validity and reliability of the questionnaire will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in research to accept
* Mini-Mental Test score more than or equal 24
* Previously receiving physical therapy through telerehabilitation

Exclusion Criteria:

* Any visual, hearing, and perception problems that may affect the answering the questionnaire items.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurological patients receiving physiotherapy and rehabilitation via telerehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Telerehabilitation Satisfaction Questionnaire in patients with Neurological disease | One week
  Patients get a minimum of 0 points (best condition) and a maximum of 4 points (worst condition) for each question on this scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yip MP, Chang AM, Chan J, MacKenzie AE. Development of the Telemedicine Satisfaction Questionnaire to evaluate patient satisfaction with telemedicine: a preliminary study. J Telemed Telecare. 2003;9(1):46-50. doi: 10.1258/135763303321159693. PMID 12641893